CLINICAL TRIAL: NCT06323668
Title: Cardiac Implantable Electronic Device RemOval Versus Full CoUrse Medical Treatment - the CIEDOUT Study - a Randomized Clinical Trial
Brief Title: Cardiac Implantable Electronic Device RemOval Versus Full CoUrse Medical Treatment
Acronym: CIEDOUT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Emil Loldrup Fosbol, Professor, MD, PhD, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H-23067693
Record Dates: First submitted 2024-03-07; First posted 2024-03-21 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-10

CONDITIONS: Cardiac Implantable Electronic Device Infection
Keywords: Cardiac Implantable Electronic Device; CIED; Pacemaker; Implantable cardioverter defibrillator; ICD; Possible CIED infection; Valvular endocarditis; Bacteremia; CIED extraction; Antibiotic therapy
MeSH Terms: conditions — Bacteremia

STUDY DESIGN:
Intervention Model Description: Randomized open label trial
Masking Description: None (Open Label)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cardiac implantable electronic device removal + empirical antibiotic therapy (Experimental): CIED removal + guideline antibiotic therapy (at least 10 days iv antibiotic therapy and then per oral treatment to 6 weeks total by POET criteria).
  The antibiotic therapy is targeted according to microbiological analyses per microorganism.
  The CIED removal will be done as soon as possible within 7 days.
  Interventions: Procedure: Cardiac implantable electronic device extraction
- Empirical antibiotic therapy (No Intervention): Guideline antibiotic therapy (at least 10 days iv antibiotic therapy and then per oral treatment to 6 weeks total by POET criteria). The antibiotic therapy is targeted according to microbiological analyses per microorganism.

INTERVENTIONS:
Procedure: Cardiac implantable electronic device extraction — The CIED removal will be done as soon as possible within 7 days.
  Arms: Cardiac implantable electronic device removal + empirical antibiotic therapy

SUMMARY:
The CIEDOUT study is an open label randomized trial in patients with possible cardiac implantable electronic device (CIED) infection.

The hypothesis is that CIED removal + guideline antibiotic therapy is better than 6-weeks antibiotic therapy alone in preventing death or relapse of bacteremia in patients with bacteremia and possible CIED infection (not definite CIED infection).

The objective of this study is to test whether CIED removal + guideline antibiotic therapy is superior to 6-weeks antibiotic therapy alone in prevention of the composite endpoint of death or relapse bacteremia after 6 months of follow-up in patients with CIED and systemic infection but without definite CIED infection.

DETAILED DESCRIPTION:
Complete removal of cardiac implantable electronic devices (CIEDs) is recommended for all patients with confirmed CIED infection under initial empirical antibiotic therapy by guidelines. However, the current 2023 European Society of Cardiology (ESC) guidelines on treatment of possible CIED infection are mostly based on expert opinions and/or observational studies. No previous randomized clinical trial has been conducted, why the CIEDOUT study is the first randomized clinical trial with high evidence investigating treatment of possible CIED infections. The CIEDOUT study will affect future clinical guidelines and optimize treatment and prognosis for future patients with possible CIED infection.

The hypothesis is that CIED removal + guideline antibiotic therapy is superior to 6-weeks antibiotic therapy alone in preventing death or relapse of bacteremia in patients with bacteremia and possible CIED infection (not definite CIED infection). The investigators want to test whether CIED removal + guideline antibiotic therapy is superior to 6-weeks antibiotic therapy in prevention of the composite endpoint of death or relapse bacteremia after 6 months of follow-up in patients with CIED and systemic infection but without definite CIED infection.

The study is a randomized open label trial. Patients will be allocated by 1:1 randomization to CIED extraction + guideline antibiotic therapy or 6-weeks antibiotic therapy alone. The primary outcome is a composite endpoint of death or relapse bacteremia (same microorganism) within 6 months after randomization. The secondary outcomes are days alive and out-of-hospital to 6 months, death, readmission for any cause, device extraction, relapse of bacteremia (the same microorganism), relapse of bacteremia (all species), and definite CIED infection.

All patients suspected of CIED infection or patients with bacteremia + CIED will be screened for inclusion in the CIEDOUT study according to the ESC modified diagnosis criteria. To enable timely identification of possible candidates, a surveillance system will be set up combining data from The Danish Pacemaker and implantable cardioverter-defibrillator (ICD) registry and then real-time bacteremia surveillance data through The Danish nationwide clinical Microbiology Database (MiBa). Hence, whenever a relevant bacteremia is identified, the CIED registry will then by queried for whether that patient also has CIED. Randomization allocation ratio is 1:1 through a computerized application via RedCap. Patients will be entered into the "intention to treat" analysis.

The patients will be randomized to CIED removal and/or medical therapy (at least 10 days iv antibiotic therapy and then per oral treatment to 6 weeks total by POET criteria). The CIED removal will be done as soon as possible within 7 days. The study-outcomes will be assessed at three routine clinical check-ups as part of the standard treatment at 1 week, 4 weeks, and 3 months after randomization. Within 6 months after randomization, patients will be followed for outcomes through medical charts and the national health registries. After that, the patients will be assessed for outcomes on an annual basis by medical chart review and the Danish nationwide registries.

The total trial duration is expected to be 14 years. Inclusion period for the main paper is expected to be 4 years and then follow-up for 3 months for the last included patients. Hereafter, patients will be followed for outcomes annually through medical charts and the national health registries up to 10 years after the last included patient until 2038.

Based on prior studies and especially preliminary data, it is estimated that approximately 29% of patients will experience a primary event by 6 months in the medical treatment group and 12% in the extraction group. In order to have 80% power to detect difference in total primary endpoints between the treatment groups, at least 174 patients will be needed (87 in each study arm) over a median follow-up of 3 years to be able to reject the null hypothesis with a power of 80% and a risk of type I error of 5. Assuming a steady rate of patients with the inclusion criteria, there will be approximately 100 incident cases available for the CIEDOUT study annually in Eastern Denmark based on preliminary data. If 60% of these consent to the study, 60 incident patients per year will be included. By 3 years, 180 incident patients will then be included.

ELIGIBILITY:
Inclusion Criteria:

Possible CIED infection*

AND

Bacteremia/fungemia with S. aureus detected in ≥1 positive blood culture(s) or CoNS, Cutibacterium spp., Candida spp, Streptococcus spp. (except Streptococcus pneumoniae), and Enterococcus faecalis detected in ≥2 positive blood cultures.

OR

Left-sided valve infective endocarditis

AND

Possible CIED infection*

AND

Bacteremia/fungemia detected in ≥1 positive blood culture(s) with S. aureus, CoNS, Cutibacterium spp., Candida spp., Streptococcus spp. (except Streptococcus pneumoniae), and Enterococcus faecalis

Exclusion Criteria:

* Unavailable for follow-up (e.g. tourist)
* Unwilling to sign informed consent
* Unable to sign informed consent

OR

At least one of the following criteria

* Not a candidate by clinician discretion
* Definite CIED infection*
* Clinical frailty score ≥7
* EUROSCORE II >33%
* Forced expiratory volume in one second (FEV1) <1L or <30% of expected

  * By the modified Duke and ESC diagnostic criteria

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2024-05-17 (Actual); Primary Completion 2028-06 (Estimated); Study Completion 2038-01-31 (Estimated)

PRIMARY OUTCOMES:
Rate of death or relapse bacteremia | 6 months after randomization
  Composite endpoint of death or relapse bacteremia (same microorganism)

SECONDARY OUTCOMES:
Days alive and out-of-hospital | 6 months after randomization
Rate of death | 6 months after randomization
Rate of readmission for any cause | 6 months after randomization
Rate of cardiac implantable electronic device extraction | 6 months after randomization
  First CIED extraction for the medical group and second for the extraction group
Rate of relapse bacteremia (the same microorganism) | 6 months after randomization
Rate of bacteremia (all species) | 6 months after randomization
Rate of definite CIED infection | 6 months after randomization

CONTACTS AND LOCATIONS:
Overall Officials: Emil L Fosbøl, MD, PhD, Principal Investigator — Department of Cardiology, Copenhagen University Hospital, Rigshospitalet
Locations (1):
- Copenhagen University Hospital, Rigshospitalet, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No